CLINICAL TRIAL: NCT05382091
Title: A Phase II Multi-Center Safety Study Examining the Use of the O'Neil Long Acting Naltrexone Implant (OLANI) in Opioid Dependent Persons Receiving Repeat Dosing
Brief Title: Evaluation of the O'Neil Long Acting Naltrexone Implant in Opioid Dependent Persons
Acronym: GM0020
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Go Medical Industries Pty Ltd (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); New York State Psychiatric Institute (Other); Columbia University (Other); The Emmes Company, LLC (Industry); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM0020; 4UH3DA047720-03 (NIH); 240359 (Other: NIH ERA Human Subjects Study Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: naltrexone; opioids; OLANI implant; opioid use disorder; opioid dependence; opioid receptor antagonist
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OLANI (naltrexone implant) (Experimental): 2 OLANI implants containing 60% naltrexone (3.6 g total NXT) administered at Day 0 with repeat dosing of a single implant at Week 13 (within a window of 12-16 weeks). The repeat single dosing may be repeated 3 times in total.
  Interventions: Drug: naltrexone implant

INTERVENTIONS:
Drug: naltrexone implant — 3.6 g per implant set each containing 60% naltrexone
  Other Names: OLANI; O'Neil Long Acting Naltrexone Implant

SUMMARY:
This study will examine the safety and efficacy of the O'Neil Long Acting Naltrexone Implant (OLANI) in persons with opioid dependency who are seeking relapse-prevention treatment. All participants will be treated in an open label manner. No randomization will occur. The OLANI is a long-acting biodegradable form of naltrexone which is implanted in the abdominal region. It is hypothesized that the OLANI will produce blood levels sufficient to block the effects of opioids for an extended period allowing patients to engage in psychosocial treatment and recovery over the long term. After the initial set of implants, participants will be offered 3 sets of single implants 13 weeks, each with an acceptable window of 12-16 weeks after the previous dose.

DETAILED DESCRIPTION:
This is a Phase II, multi-center, open-label study designed to evaluate the safety profile and the efficacy of the OLANI when used in participants who meet the diagnosis of opioid use disorder (OUD), as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), and who will be voluntarily seeking relapse-prevention treatment using the naltrexone (NTX) implant.

Participants eligible for the study have diagnosed OUD, have completed withdrawal from opioids, and are no longer physically dependent at the time of study enrollment. After completing the informed consent process for the study, all participants will receive their initial OLANI set (two implants) implanted subcutaneously by a study surgeon and will be followed by a medical and surgical research team, receiving medical management intervention and blood draws to measure levels of NTX and its metabolite, 6-beta-naltrexol (6BN).

For interested participants, a standard dose of OLANI (standard dose contains 1 x OLANI, for a total of 1.8 g NTX) will be offered 13 weeks (91 days), within an acceptable dosing window of 12-16 weeks (84-112 days) after the initial loading dose, with a preference for participants to receive the dose between 84-91 days. Participants will continue to be offered a repeat standard dose of OLANI every 13 weeks (91 days), within an acceptable dosing window of 12-16 weeks (84-112 days) after their previous dose for a further two repeats. This will result in a maximum of 4 procedures within 36 to 48-weeks. All participants will be followed up until 60 weeks post their initial IP procedure, irrespective of the number of procedures that they have. This will result in a total study duration of 60 weeks for all participants.

ELIGIBILITY:
Inclusion Criteria:

* All genders between 18 and 65 (inclusive) years old
* Meet criteria for a current (within the previous 12-months) DSM-5 diagnosis of OUD at screening, and voluntarily seeking relapse-prevention treatment with NTX implant
* Completed opioid withdrawal as demonstrated by a negative naloxone challenge test (i.e., has tolerated naloxone 0.8 mg)
* Individuals currently treated with NTX will be eligible to receive the implant at the end of the dosing interval of either Vivitrol or oral NTX
* Have no medical or psychiatric contraindications to treatment either with NTX or with the OLANI, as determined by the site clinician and based on medical history and current health status
* Able to sufficiently speak and understand English and understand study procedures
* Able and willing to provide written informed consent
* Able and willing to provide detailed contact information for both self and for close contact(s) on the locator form
* Able and willing to comply with the requirements and procedures of the protocol, including tolerating a minor surgical procedure with local anesthetic for placement of the implant sets into the subcutaneous tissue of the abdomen
* Have an initial weight between 45.3 and 130 kg (inclusive) or have a BMI of 18.5 to 35.0 (inclusive)
* For female participants of childbearing potential, a willingness to practice an effective method of birth control for the duration of participation in the study. Acceptable methods of birth control are specified on the data collection form and in the Manual of Procedures (MOP), and methods other than those specified are not permitted, except in combination with a study-acceptable method; and willingness to complete urine pregnancy testing to confirm non-pregnant status, as per the study schedule and as requested by the site clinician.

Exclusion Criteria:

* Has a condition, disease state, previous medical history, or observed abnormality(ies) (including physical examination, electrocardiogram [ECG], laboratory evaluation, or urinalysis finding) identified during screening that, in the opinion of the site clinician, would preclude safe participation in the study, would affect the ability of the participant to adhere to the protocol, or would interfere with the study assessments, including, but not limited to the following:

  * A significant neurological (including cognitive and psychiatric disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable using protocol-allowed medication(s) for the 30 days immediately preceding the proposed administration of OLANI
  * Has had significant suicidal ideation or behavior within the past year
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value more than three times the upper limit of normal, or a different indicator of clinically significant liver cirrhosis (e.g., bilirubin and albumin will also be assessed)
  * Has a condition (e.g., chronic pain) that requires ongoing treatment with opiate based medication
  * Has any contraindicated medical condition per the approved labelling for NTX containing products
* Has physiological dependence on alcohol and/or sedative-hypnotics that require medical detoxification
* If female, is currently pregnant or breastfeeding, is planning to conceive during the period of study engagement, has a positive blood pregnancy test, or is unwilling to practice effective contraception during study participation
* Has received a NTX implant in the last 12 months
* Has a known hypersensitivity to NTX
* Is not able to provide blood samples due to extensive vein damage
* Has a known hypersensitivity to polylactic acid based materials, including disposable sutures or implants
* Has a known hypersensitivity to local anesthesia
* Is prone to skin rashes, skin irritation, or has a diagnosed or observed skin condition (e.g., recurrent eczema)
* Is tattooed in the proposed implantation area or demonstrates any abnormal skin tissue in the proposed implantation area
* Currently confined or detained in a penal institution or sentenced to such an institution under a criminal or civil statute or detained in other facilities by virtue of statutes.
* Any additional condition(s) that, in the investigator's opinion, would prohibit the participant from completing the study or that would not be in the best interest of the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | time from from placement of first implant set until end of study at 60 weeks.
  Incidence and Severity of TEAEs
Adverse Events of Special Interest (AESI) | time from from placement of first implant set until end of study at 60 weeks.
  Incidence of AESIs related to the surgical procedure and local reaction to the implant over time
Deaths | time from from placement of first implant set until end of study at 60 weeks.
  Incidence of study deaths
Serious Adverse Events (SAEs) | time from from placement of first implant set until end of study at 60 weeks.
  Incidence of SAEs
Adverse events (AEs) causing study discontinuation | time from from placement of first implant set until end of study at 60 weeks.
  AEs that lead to study discontinuation
Opioid overdose events | time from from placement of first implant set until end of study at 60 weeks.
  Incidence of opioid overdose events
Laboratory abnormalities | time from from placement of first implant set until end of study at 60 weeks.
  Incidence and Severity of lab abnormalities
Suicidality | time from from placement of first implant set until end of study at 60 weeks.
  incidence of suicidal ideation and suicidal behavior captured with the Columbia-Suicide Severity Rating Scale (C-SSRS)
Concomitant medications | time from from placement of first implant set until end of study at 60 weeks.
  Proportion of participants who initiate concomitant medications

SECONDARY OUTCOMES:
AUC0-t of naltrexone | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  area under the plasma concentration-time curve from 0 to the time of last measurable concentration (AUC0-t)
AUC0-t of 6-beta-naltrexol | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  area under the plasma concentration-time curve from 0 to the time of last measurable concentration (AUC0-t)
AUC0-infinity of naltrexone | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  area under the plasma concentration-time curve extrapolated to infinity (AUC0-infinity)
AUC0-infinity of 6-beta-naltrexol | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  area under the plasma concentration-time curve extrapolated to infinity (AUC0-infinity)
Cmax of naltrexone | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  Single-dose pharmacokinetic (PK) measurement of the plasma naltrexone concentration (Cmax) after dosing on Day 1
Cmax of 6-beta-naltrexol | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  Single-dose PK measurement of the plasma 6-beta-naltrexol concentration (Cmax) after dosing on Day 1
Tmax of naltrexone | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  Single-dose PK measurement of the time to reach the maximum plasma naltrexone concentration (Tmax) after dosing on Day 1
Tmax of 6-beta-naltrexol | collected before each implant administration (pre-dose), and 3 hours, 7 days, 14 days, 28 days, then every 14 days until next implant procedure. PK sampling is reduced to every 28 days after 12 weeks if the next implant procedure is not completed.
  Single-dose PK measurement of the time to reach the maximum plasma naltrexone concentration (Tmax) after dosing on Day 1
Proportion of participants that maintain a minimum plasma concentration | up to Week 60
  Proportion of participants who maintain NTX blood levels of ≥2 ng/mL
Proportion of participants that maintain a minimum plasma concentration | up to Week 60
  Proportion of participants who maintain NTX blood levels of ≥1.16 ng/mL
Abstinence from drugs of abuse by UDS | pre-dose (prior to each implant procedure) and at every study visit through Week 60.
  Proportion of participants who maintain abstinence from opioids, benzodiazepines; barbiturates; cocaine; amphetamine; methamphetamine; phencyclidine (PCP); ecstasy (MDMA); and marijuana (THC) as measured through a urine drug screen (UDS)
Abstinence from drugs of abuse by Timeline Followback (TLFB) | At every study visit through Week 60 except for days of implant procedures.
  Proportion of participants who maintain abstinence from opioids, benzodiazepines; barbiturates; cocaine; amphetamine; methamphetamine; phencyclidine (PCP); ecstasy (MDMA); and marijuana (THC) as measured through a urine drug screen (UDS)
Abstinence from alcohol | pre-dose (prior to each implant procedure) and at every study visit through Week 60.
  Proportion of participants who maintain abstinence from alcohol as measured using and alcohol breathalyzer
Opioid craving (VAS) | pre-dose (prior to each implant procedure) and at every study visit through Week 60.
  The craving for opioids will be measured using a horizontal visual analog scale (VAS), which ranges from 0 (no craving) to 10 (most intense craving possible).
Opioid withdrawal (SOWS) | pre-dose (prior to each implant procedure) and at every study visit through Week 60.
  The SOWS is a 16-item questionnaire designed to measure the severity of opioid withdrawal symptoms. The participant rates the intensity of symptoms using a 5-point scale; with 0 representing "not at all" and 4 representing "extremely".
Opioid withdrawal (COWS) | pre-dose (prior to each implant procedure) and at every study visit through Week 60.
  The COWS is a questionnaire designed to measure 11 common opioid withdrawal signs and symptoms. The summed score provides information about the severity of opioid withdrawal and the level of physical dependence on opioids. Total scores range from 0 to 47, and withdrawal is classified as mild (5-12), moderate (13-24), moderately severe (25-36), or severe (>36)
Hamilton Depression Rating Scale (HDRS) | At every study visit through Week 60 except for days of implant procedures.
  Assessment of Depression/Mood via the HDRS, is a clinician-administered instrument, useful for following both depression and suicidal ideation, and for following typical symptoms of subacute withdrawal (e.g., low appetite, fatigue, poor sleep). A score of 1 or more to item 3 (suicidality) prompts a clinician assessment for suicide risk before leaving the clinic.
Brief Symptom Inventory 18 (BSI-18) | Baseline, Day 28, Day 42, Day 56, Day 84, and then every 28 days until Week 60.
  Assessment of Depression/Mood via the BSI-18; comprising 18 items (ranging from 0 = not at all to 4 = extremely), assesses psychiatric symptoms in three distinct domains: depression, anxiety, and somatization. The total score ranges from 0 to 72 with higher scores indicating higher symptom severity.
Quality of Life Score (QoL) | Day 28, Day 42, Day 56, Day 84, and then every 28 days until Week 60.
  Quality of life as measured through Quality of Life Enjoyment and Satisfaction Questionnaire (short form). is a 16 item self-administered questionnaire that captures life satisfaction over the past week. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). Scores from the individual items are added together and reported as percentage maximum possible score. The Total Score is reported as percentage maximum possible % Max = Raw-minimum score/maximum score-minimum score. (Raw score minus the minimum possible raw score divided by the maximum possible raw score minus the minimum possible raw score). If items are left blank the maximum and minimum scores must be modified to reflect the number of items scored.
Treatment Satisfaction (TSQM-14) | Repeat implant procedure days and at Week 60.
  The TSQM-14 is comprised of 14 questions that provide scores on four scales: effectiveness (3 items), side effects (5 items), convenience (3 items) and global satisfaction (3 items). With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — New York State Psychiatric Institute

IPD SHARING:
Plan to Share IPD: No